CLINICAL TRIAL: NCT05322070
Title: Phase 4 Study of YUTIQ® (Fluocinolone Acetonide Intravitreal Implant) 0.18 mg in the Treatment of Chronic Non-Infectious Posterior Segment Uveitis (Intraocular Inflammation Study)
Brief Title: Fluocinolone Acetonide Intravitreal Implant 0.18 mg in the Treatment of Chronic Non-Infectious Posterior Segment Uveitis
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Alimera Sciences (Industry)
Collaborators: CBCC Global Research (Network)
Responsible Party: Sponsor
Organization: ANI Pharmaceuticals (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EYP-YUT-002
Record Dates: First submitted 2022-03-02; First posted 2022-04-11 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Uveitis, Posterior
Keywords: Intraocular Inflammation; Fluocinolone Acetonide Intravitreal Implant
MeSH Terms: conditions — Uveitis, Posterior; Uveitis | interventions — Fluocinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Fluocinolone Acetonide 0.18 mg (Experimental): Fluocinolone Acetonide Intravitreal Implant 0.18 mg
  Interventions: Drug: Fluocinolone Acetonide Intravitreal Implant 0.18 mg

INTERVENTIONS:
Drug: Fluocinolone Acetonide Intravitreal Implant 0.18 mg — YUTIQ® 0.18 mg as an intravitreal injection in the designated study eye.
  Other Names: YUTIQ 0.18 mg

SUMMARY:
A study to evaluate the safety and efficacy of YUTIQ® 0.18 mg intravitreal implant for the management of chronic non-infectious posterior segment uveitis (intraocular inflammation) that has responded to previous steroid therapy.

DETAILED DESCRIPTION:
This is a prospective, phase 4, open-label, uncontrolled, 2-year follow-up study to evaluate the safety and efficacy of YUTIQ® (fluocinolone acetonide intravitreal implant) 0.18 mg for the management of chronic non-infectious posterior segment uveitis (intraocular inflammation) that has responded to previous steroid therapy. Patients will receive YUTIQ® 0.18 mg as an intravitreal injection in the designated study eye and will be followed for 24 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female in good general health at least 18 years of age at time of consent.
* Presence of active, recurrent, unilateral or bilateral non-infectious uveitis affecting the posterior segment (intraocular inflammation) with a duration of at least 3 months from initial diagnosis, as determined by the Investigator. Intermediate or panuveitis will also be allowed if posterior segment involvement is part of the diagnosis.
* Posterior segment inflammation that has previously demonstrated a clinical response to ≥1 localized corticosteroid treatment (eg, topical steroid 2 to 4 times per day or intra- or peri-ocular injection).
* Presence of macular edema as measured by spectral-domain - optical coherence tomography (SD-OCT) (≥325 microns on Heidelberg SPECTRALIS and ≥315 microns on Zeiss CIRRUS).
* Best corrected visual acuity (BCVA) of the study eye 35-75 letters on the ETDRS chart (Snellen range 20/30 to 20/200).
* Not planning to undergo elective ocular surgery during the study.
* Able to understand, sign the Informed Consent Form (ICF).
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* History of macular edema due to diabetes, retinal vein occlusion (RVO), age-related macular degeneration (AMD), or any non-inflammatory cause.
* Intraocular inflammation with infectious etiology.
* Diagnosis of uncontrolled glaucoma or ocular hypertension at Screening, unless study eye is being treated with ≤2 intraocular pressure (IOP)-lowering medications and/or has been previously treated with an incisional surgical procedure OR glaucoma laser procedure resulting in stable IOP in the normal range (10 to 21 mmHg).
* Intraocular pressure >21 mmHg or concurrent therapy at Screening with >2 IOP-lowering pharmacologic agents in the study eye.
* Ocular malignancy in either eye, including choroidal melanoma.
* Previous viral retinitis.
* Toxoplasmosis scar or scar related to previous viral retinitis in the study eye.
* Ocular and periocular infections such as diseases of the cornea and conjunctiva including epithelial herpes simplex keratitis (dendritic keratitis), vaccinia, and varicella, mycobacterial infections of the eye, or fungal diseases of ocular structures.
* Hypersensitivity to any of the ingredients contained in YUTIQ®.
* Media opacity precluding evaluation of retina and vitreous (eg, vitreous hemorrhage).
* Any current retinal detachment or retinoschisis in insertion in the study eye.
* Chronic hypotony, defined as <6 mmHg for at least 1 month's duration, and documented on at least two separate visits.
* Ocular surgery within 12 weeks prior to Day 1.
* YAG laser capsulotomy within 30 days prior to Day 1.
* Prior intravitreal treatment with Retisert®, ILUVIEN®, or YUTIQ® (0.18 mg) within 36 months prior to Day 1.
* Prior intravitreal treatment with OZURDEX® within 12 weeks prior to Day 1.
* Prior intravitreal treatment with Triesence® or TRIVARIS™ (triamcinolone) within 12 weeks prior to Day 1.
* Peri-ocular or subtenon steroid treatment within 12 weeks prior to Day 1.
* Radiation to the head or neck within 2 years prior to Screening.
* Steroid allergy, particularly to fluocinolone.
* Any systemic condition that requires chronic systemic anti-inflammatory, steroid, or immunosuppressive therapy (subjects on a stable dose of oral prednisone <7.5 mg per day for a non-ocular indication may be included).
* Positive test for human immunodeficiency virus (HIV), tuberculosis, or syphilis in the past 2 years or during Screening.
* Any severe acute or chronic medical (eg, cancer diagnosis) or psychiatric condition that could increase the risk associated with study participation or could interfere with the interpretation of study results and make the subject inappropriate for study enrollment.
* Any other systemic or ocular condition which, in the judgment of the Investigator, could make the subject inappropriate for study enrollment.
* Treatment with an investigational drug or device within 30 days prior to Day 1.
* Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of contraception as outlined in the protocol from at least 14 days prior to Day 1 until the final study visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in BCVA | Month 6
  • Mean change from baseline in BCVA letter score in the study eye measured by EDTRS.
Change in CST | Month 6
  • Mean change from baseline central subfield thickness (CST, also known as central foveal thickness) measured by SD-OCT in the study eye.

SECONDARY OUTCOMES:
Recurrence of non-infectious inflammation | Months 1, 3, 6, 12, 18, and 24
  • Time to recurrence of non-infectious inflammation in the study eye defined as an increase in CST.
Presence of vascular leakage | Months 1, 3, 6, 12, 18, and 24.
  • Presence of vascular leakage as measured by wide field fluorescein angiography.
Resolution of macular edema | Months 1, 3, 6, 12, 18, and 24
  • Proportion of subjects with resolution of macular edema (central subfield thickness CST) as measured by SD OCT.
Change in BCVA letter score | Day 14 and at Months 1, 3, 12, 18, and 24
  • Mean change from baseline in BCVA letter score in the study eye measured by EDTRS.
Change from baseline in CST | Months 1, 3, 12, 18, and 24
  • Mean change from baseline in CST measured by SD-OCT in the study eye.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cutino, Study Chair — Alimera Sciences Inc
Locations (23):
- United States (23):
  - Retina Consultants of Orange County, Fullerton, California
  - Macula and Retina Institute, Glendale, California
  - California Eye Specialists Medical Group, Pasadena, California
  - Retinal Consultants Medical Group, Sacramento, California
  - Retina Associates of Colorado, Lakewood, Colorado
  - Advanced Research, Coral Springs, Florida
  - Retina Specialists of Tampa, Wesley Chapel, Florida
  - Marietta Eye Clinic, Marietta, Georgia
  - Retinal Vitreal Consultants Ltd., Chicago, Illinois
  - Illinois Retina Associates, S.C., Oak Park, Illinois
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Opthalmic Consultants of Boston, Boston, Massachusetts
  - Massachusets Eye Research and Surgery Institution, Waltham, Massachusetts
  - Foundation for Vision Research, Grand Rapids, Michigan
  - Midwest Vision Research Foundation at Pepose Vision Institute, Chesterfield, Missouri
  - Retina Consultants, Fargo, North Dakota
  - Retina Vitreous Associates, Toledo, Ohio
  - Erie Retina Research, LLC, Erie, Pennsylvania
  - Tennessee Retina, Nashville, Tennessee
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Consultants of Texas, Katy, Texas
  - Valley Retina Institute, PA, McAllen, Texas
  - Medical Center Opthalmology Associates, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No